CLINICAL TRIAL: NCT06608355
Title: A Phase I Study to Assess the Safety, Tolerability and Preliminary Efficacy of NouvNeu001 Injection in the Treatment of Early-onset Parkinson's Disease
Brief Title: The Safety, Tolerability and Preliminary Efficacy of NouvNeu001 for Early-onset Parkinson's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: iRegene Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NouvNeu001-03
Record Dates: First submitted 2024-09-14; First posted 2024-09-23 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-09

CONDITIONS: Early-onset Parkinson's Disease
Keywords: Early-onset Parkinson's Disease; Dopaminergic Progenitor Cells
MeSH Terms: conditions — Parkinsonian Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- NouvNeu001 (Experimental)
  Interventions: Biological: Human Dopaminergic Progenitor Cells

INTERVENTIONS:
Biological: Human Dopaminergic Progenitor Cells — Single injection of Human Dopaminergic Progenitor Cells into the putamen of brain.

SUMMARY:
The goal of this clinical trial is to learn about the safety of NouvNeu001 injection in Early-onset Parkinson's Disease (EOPD) patients. It will also learn about the effects of NouvNeu001 treatment. The main questions it aims to answer are:

What medical problems do participants have when transplanting NouvNeu001 into bilateral putamen using stereotactic neurosurgery? Does injection of NouvNeu001 improve the motor function and non-motor function in participants?

Participants will:

Be injectioned the NouvNeu001 into bilateral putamen using stereotactic neurosurgery.

Take immunosuppressants to prevent potential immune rejection for 24 to 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old, male or female
* Able to understand the rationale of the clinical trial and sign informed consent form (ICF)
* Diagnosis of Early-onset Parkinson's Disease in accordance with the MDS clinical diagnostic criteria for Parkinson's disease, and the age of onset was ≤50 years old
* Medically suitable for neurosurgery under anesthesia and able to participate in Computed Tomography (CT)/Magnetic Resonance Imaging (MRI) scan.
* Hoehn-Yahr staging for "off" episodes is 2 to 4
* The MDS-UPDRS-III score in the "off" state >30, and positive for the Acute Levodopa Challenge Test (ALCT)
* Acceptable laboratory test results during screening and prior to transplantation

Exclusion Criteria:

* Atypical Parkinsonism
* Patients who have had previous pallidotomy, striatal or extrapyramidal surgery or other brain surgery; as well as other surgical procedures that are judged by the investigator to affect patient's participation in this study; Patients with surgical contraindications or other neurosurgical contraindications
* Patients who have a previous head CT/MRI examination showing cerebral trauma, vascular malformation, hydrocephalus, brain tumor, etc., and patients who have brain imaging abnormalities in the striatum or other brain areas leading to a significantly increased risk for surgery
* Patients with a history of severe cardiovascular and cerebrovascular diseases
* Patients with a history of malignant tumors
* Patients who have received stem cell therapy for Parkinson's disease within 2 years before signing the ICF
* Patients with active disseminated intravascular coagulation and significant hemorrhagic tendency within 3 months prior to screening, or who cannot temporarily suspend anti-platelet agents or other anti-coagulant medications for at least 5 days before surgery
* Patients with long-term, heavy use of glucocorticoids or immunosuppressive drugs within 3 months prior to signing the ICF
* Patients with a history of mental illness who are deemed unfit to participate in the study by the investigator; or a history of suicidal ideation or suicide attempts within the past year or currently
* Patients who have used botulinum toxin within 6 months prior to signing the ICF
* Patients with active epilepsy or currently on anti-epileptic drugs
* Patients with a history of dementia or severe cognitive disorder, or the score of MDS-UPDRS 1.1 during screening is > 3; poor compliance, inability to accurately keep diary, and/or inability to sign ICF due to dementia
* Patients with severe depression or with severe anxiety
* Patients with the following abnormalities during screening, including: Abnormal coagulation; Abnormal immunological tests, and assessed by the investigator it is not suitable to participate in the trial; Hypertensive patients with poorly controlled blood pressure and patients with severe postural hypotension; Diabetic patients with poorly controlled blood glucose
* Patients with other combined severe systemic diseases, such as pulmonary heart disease, moderate to severe asthma, severe chronic obstructive pulmonary disease (COPD)
* Presence of one of the following: positive for human immunodeficiency virus (HIV) antibody, treponema pallidum antibody, hepatitis C virus (HCV) antibody and HCV RNA; Hepatitis B virus (HBV) surface antigen positive and HBV DNA copy number > detection of normal values; Tuberculosis is in the active stage; Other active infections that the investigator believes may affect Patients' participation in the study or affect study outcomes
* Patients with alcohol addiction or positive for drug of abuse testing
* Patients with a history of contraindication or allergy to the drugs used during the study or any of its components, or are allergic to the same drugs or other macrolides, or have allergies
* Female of childbearing potential who are not surgically sterilized/premenopausal/unwilling to use medically approved effective contraception with 2 years after administration of investigational drug and lactating women; men who are not surgically sterilized/unwilling to use medically approved effective contraception with 2 years after administration of investigational drug
* Patients who have received electric shock therapy within 30 days prior to surgery
* Patients who are participating in other clinical trials, or have been enrolled in other clinical studies and received intervention therapy within 3 months prior to the surgery
* Patients with poor compliance based on clinical evaluation of the investigator
* Patients who are being treated with drugs such as apomorphine, or levodopa/carbidopa infusion therapy
* Patients with severe dyskinesia in both on- and off-drug states

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Enrollment to 96 weeks post-transplant.
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs).

SECONDARY OUTCOMES:
The Motor Function and Non-motor Function | Baseline to 48 weeks and 96 weeks post-transplant
  Changes in Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part I-IV Score from baseline. A higher score indicates more severe symptoms or worse health.

OTHER OUTCOMES:
Positron Emission Tomography Imaging | Baseline to 48 weeks post-transplant.
  Change in uptake value from baseline using positron emission tomography (PET).
Dopamine Metabolism | Baseline to 48 weeks post-transplant.
  Change in the levels of dopamine and its metabolites from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College Hust, Wuhan, Hubei, China